CLINICAL TRIAL: NCT04717180
Title: Post Stroke Aphasia Rehabilitation Using Computer-based Arabic Software Program: A Randomized Control Trial
Acronym: aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: aphasia software
Record Dates: First submitted 2021-01-02; First posted 2021-01-22 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2020-12

CONDITIONS: Aphasia Rehabilitation
Keywords: aphasia, post stroke
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group I (Active Comparator): patients who received rehabilitation using the software program for aphasia rehabilitation
  Interventions: Behavioral: aphasia rehabilitation using software program or conventional therapy
- group II (Active Comparator): patients who received rehabilitation using the conventional therapy
  Interventions: Behavioral: aphasia rehabilitation using software program or conventional therapy

INTERVENTIONS:
Behavioral: aphasia rehabilitation using software program or conventional therapy — Patients were randomized into two groups: group I who received therapy using the software aphasia rehabilitation program and group II who received conventional (traditional) language therapy
  Other Names: aphasia rehabilitation using the conventional language therapy

SUMMARY:
Aphasia is a disorder of language processing caused by a lesion in particular brain regions. Treatment aims at improving or restoring impaired function or at compensating for deficits. More recently, computer technology has been integrated into treatment options. In this study, a detailed and comprehensive computerized software program for aphasia rehabilitation is designed for the treatment of Arabic speaking Egyptian aphasic patients.

Aim of the study: design a computerized software program for the rehabilitation of Arabic speaking Egyptian aphasic patients.

DETAILED DESCRIPTION:
Aphasia is a disorder of language processing caused by a lesion in particular brain regions. Treatment aims at improving or restoring impaired function or at compensating for deficits. More recently, computer technology has been integrated into treatment options. In this study, a detailed and comprehensive computerized software program for aphasia rehabilitation is designed for the treatment of Arabic speaking Egyptian aphasic patients.

Aim of the study: design a computerized software program for the rehabilitation of Arabic speaking Egyptian aphasic patients.

Subjects: The study was conducted on 50 patients with aphasia who attend the unit of Phoniatrics during the period of one year, Department of Otorhinolaryngology, Alexandria Main University Hospitals.

Methodology: The training materials were designed as a software program. Each patient was subjected to assessment before and after the application of the rehabilitation program. Patients were randomized into two groups: group I who received therapy using the software aphasia rehabilitation program and group II who received conventional (traditional) language therapy. Therapy continued for 48 sessions over six months.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of aphasia
* Age 18 years or more

Exclusion Criteria:

* Intellectual disabilities.
* Visual impairment.
* Hearing impairment.
* Associated dysarthria and or apraxia of speech.
* Associated psychiatric disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
The primary outcome was a measure of improvement in language abilities. | 6 months
  The primary outcome was a measure of improvement in language abilities. It was measured (after 48 sessions) using Boston Diagnostic Aphasia Examination (BDAE) Arabic version to detect any significant improvement in language

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Main University Hospitals, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No